CLINICAL TRIAL: NCT02478398
Title: A Phase III, Randomized, Placebo-Controlled Clinical Trial to Study the Efficacy and Safety of MK-3641, a Ragweed (Ambrosia Artemisiifolia) Sublingual Immunotherapy Tablet, in Children With a History of Ragweed-Induced Rhinoconjunctivitis With or Without Asthma
Brief Title: Efficacy and Safety Study of RAGWITEK™ (MK-3641) in Children With Ragweed-Induced Rhinoconjunctivitis With or Without Asthma (MK-3641-008)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3641-008; 2014-004341-27 (EudraCT Number); MK-3641-008 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-06-22; First posted 2015-06-23 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Epinephrine; Albuterol; Loratadine; Olopatadine Hydrochloride; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short ragweed pollen allergen extract (Experimental): Participants receive one sublingual tablet containing 12 units of Ambrosia artemisiifolia major allergen number 1 (Amb a 1-U), once daily (QD) for up to 35 weeks. Participants may use study-provided rescue medication(s) as needed to treat rhinoconjunctivitis symptoms.
  Interventions: Biological: Short ragweed pollen allergen extract; Drug: Self-injectable epinephrine; Drug: Albuterol/Salbutamol; Drug: Loratadine; Drug: Olopatadine; Drug: Mometasone furoate monohydrate
- Placebo (Placebo Comparator): Participants receive one placebo sublingual tablet, QD for up to 35 weeks. Participants may use study-provided rescue medication(s) as needed to treat rhinoconjunctivitis symptoms.
  Interventions: Biological: Placebo; Drug: Self-injectable epinephrine; Drug: Albuterol/Salbutamol; Drug: Loratadine; Drug: Olopatadine; Drug: Mometasone furoate monohydrate

INTERVENTIONS:
Biological: Short ragweed pollen allergen extract — One sublingual tablet containing 12 units of Amb a 1-U, once daily (QD) for up to 35 weeks.
  Other Names: RAGWITEK™; MK-3641
  Arms: Short ragweed pollen allergen extract
Biological: Placebo — One placebo sublingual tablet, QD for up to 35 weeks.
  Arms: Placebo
Drug: Self-injectable epinephrine — Intramuscular (IM) injection with suggested doses of 0.15 mg for participants weighing 15-30 kg (33-66 pounds) or 0.3 mg for participants weighing ≥30 kg (≥66 pounds), as needed for severe allergic reactions. Epinephrine was only provided in countries/study sites where it was a regulatory requirement.
  Other Names: EpiPen
Drug: Albuterol/Salbutamol — Inhalation of albuterol 90 mcg/puff or salbutamol 100 mcg/puff metered dose inhaler (MDI), as needed as asthma rescue medication for those participants with asthma
  Other Names: ProAir HFA; Proventil HFA; Ventolin HFA
Drug: Loratadine — 5 mg (1 mg/mL syrup or 5 mg tablet) for participants 5 years old or 10 mg (1 mg/mL syrup or 10 mg tablet) for participants 6 to 17 years old, as needed for rhinoconjunctivitis symptoms
  Other Names: Claritin
Drug: Olopatadine — Opthalmic solution, 1 drop (0.1%) per affected eye twice daily (BID), as needed for rhinoconjunctivitis symptoms
  Other Names: Patanol
Drug: Mometasone furoate monohydrate — Intranasal spray, at doses of 1 spray (50 mcg/ spray) per nostril for participants 5 to 11 years old or 2 sprays (50 mcg/spray) per nostril for participants 12 to 17 years old, as needed for rhinoconjunctivitis symptoms
  Other Names: Nasonex

SUMMARY:
The purpose of this study is to assess the efficacy and safety of short ragweed pollen allergen extract (MK-3641, SCH 039641, RAGWITEK™) sublingual immunotherapy tablets in children aged 5 to 17 years with ragweed-induced allergic rhinitis/rhinoconjunctivitis with or without asthma. The primary hypothesis of this study is that administration of short ragweed pollen allergen extract sublingual immunotherapy tablets to children 5 to 17 years of age, compared with placebo, will result in a significant reduction in the combination of rhinoconjunctivitis symptoms and medication use over the peak ragweed season (RS).

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 4 and 17 years (inclusive) at enrollment in this study and is at least 5 years old at randomization
* Has a clinical history of significant ragweed pollen-induced allergic rhinitis/rhinoconjunctivitis of ≥1 year (at least 1 season for ages 4 to 6 years) or ≥2 years (at least 2 seasons for ages 7 to 17 years) duration diagnosed by a physician (with or without asthma) and have received treatment for the condition during the previous ragweed season
* If female, agrees to remain abstinent or use (or have their partner use) an acceptable method of birth control within the projected duration of the study.

Exclusion Criteria:

* Has a clinical history of symptomatic seasonal allergic rhinitis (and/or asthma) due to another allergen, which has required regular medication during, or potentially overlapping, the ragweed season
* Has a clinical history of significant symptomatic perennial allergic rhinitis and/or asthma due to an allergen to which the subject is regularly exposed during the ragweed season which would interfere with assessment of the treatment effect
* Has any nasal condition that could confound the efficacy or safety assessments (e.g., nasal polyposis).
* Has asthma requiring high daily doses of inhaled corticosteroids within the 6 months prior to the Screening visit
* Is either >7 years old and cannot perform reproducible FEV1 maneuvers despite coaching; OR is ≤7 years old and cannot perform reproducible FEV1 maneuvers despite coaching and has current symptoms of asthma characterized by recurrent episodes of wheezing, or episodes of cough, wheeze, difficulty in breathing, or chest tightness
* Has severe, unstable, or uncontrolled asthma, as judged by the clinical investigator, or has experienced a life-threatening asthma attack or an occurrence of any clinical deterioration of asthma that resulted in emergency treatment, hospitalization due to asthma, or treatment with systemic corticosteroids (but allowing short-acting beta agonists) at any time within the last 3 months prior to the Screening or Randomization visits
* Has a history of anaphylaxis with cardiorespiratory symptoms with prior immunotherapy, unknown cause, or inhalant allergen
* Has a diagnosis of eosinophilic esophagitis
* Has a history of chronic urticaria and/or chronic angioedema
* Has a clinical history of chronic sinusitis during the 2 years prior to the Screening or Randomization visits
* Has current severe atopic dermatitis
* Has a history of allergy, hypersensitivity, or intolerance to the ingredients of the study drug (except for Ambrosia artemisiifolia), rescue medications, or self-injectable epinephrine
* Has previously received short ragweed pollen allergen extract
* Has previously been randomized into this study
* Is participating in any other clinical study or plans to participate in another clinical study during the duration of this study

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1025 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Ellis AK, Gagnon R, Bernstein DI, Nolte H. Randomized controlled trial of ragweed sublingual immunotherapy tablet in the subpopulation of Canadian children and adolescents with allergic rhinoconjunctivitis. Allergy Asthma Clin Immunol. 2021 Dec 9;17(1):127. doi: 10.1186/s13223-021-00626-2. PMID 34886880
- [Derived] Fortescue R, Kew KM, Leung MST. Sublingual immunotherapy for asthma. Cochrane Database Syst Rev. 2020 Sep 14;9(9):CD011293. doi: 10.1002/14651858.CD011293.pub3. PMID 32926419
- [Derived] Field K, Blaiss MS. Sublingual Versus Subcutaneous Immunotherapy for Allergic Rhinitis: What Are the Important Therapeutic and Real-World Considerations? Curr Allergy Asthma Rep. 2020 Jun 16;20(9):45. doi: 10.1007/s11882-020-00934-4. PMID 32548677
- [Derived] Nolte H, Bernstein DI, Nelson HS, Ellis AK, Kleine-Tebbe J, Lu S. Efficacy and Safety of Ragweed SLIT-Tablet in Children with Allergic Rhinoconjunctivitis in a Randomized, Placebo-Controlled Trial. J Allergy Clin Immunol Pract. 2020 Jul-Aug;8(7):2322-2331.e5. doi: 10.1016/j.jaip.2020.03.041. Epub 2020 Apr 15. PMID 32304832

RESULTS

PARTICIPANT FLOW:
Groups:
- Short Ragweed Pollen Allergen Extract: Participants received one short ragweed pollen allergen extract sublingual tablet containing 12 units of Amb a 1-U, once daily (QD) for up to 35 weeks.
- Placebo: Participants received one placebo sublingual tablet, QD for up to 35 weeks.
Period: Overall Study
Arm/Group | Short Ragweed Pollen Allergen Extract | Placebo
Started | 513 | 512
Treated | 512 | 510
Completed | 461 | 491
Not Completed | 52 | 21
Not completed — Adverse Event | 20 | 5
Not completed — Lost to Follow-up | 5 | 4
Not completed — Non-Compliance With Study Drug | 5 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal By Parent/Guardian | 9 | 6
Not completed — Withdrawal By Participant | 10 | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for all treated participants.
Groups:
- Short Ragweed Pollen Allergen Extract: Participants received one short ragweed pollen allergen extract sublingual tablet containing 12 units of Amb a 1-U, QD for up to 35 weeks.
- Total: Total of all reporting groups
Arm/Group | Short Ragweed Pollen Allergen Extract | Placebo | Total
Number analyzed (Participants) | 512 | 510 | 1022
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (3.2) | 12.2 (3.1) | 12.1 (3.1)
Age, Customized [Count of Participants; unit: Participants]
  < 12 years | 206 | 204 | 410
  ≥ 12 years | 306 | 306 | 612
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 191 | 379
  Male | 324 | 319 | 643
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 18 | 14 | 32
  White | 473 | 477 | 950
  More than one race | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 21 | 36
  Not Hispanic or Latino | 490 | 483 | 973
  Not Reported | 4 | 5 | 9
  Unknown | 3 | 1 | 4
Baseline Asthma Status [Count of Participants; unit: Participants]
  Yes | 219 | 217 | 436
  No | 293 | 293 | 586

OUTCOME MEASURES:

1. Primary Outcome: Total Combined Score (TCS) During the Peak Ragweed Season (RS)
Description: TCS is daily symptom score (DSS) plus daily medication score (DMS), assessed in the peak RS (15 consecutive RS days with the highest 15-day average pollen count). The rhinoconjunctivitis (RC) DSS assesses 6 allergy symptoms measured on a scale of 0 to 3 (0=no symptoms, 3=severe symptoms; score range: 0-18). Lower DSS indicates less RC symptoms. The RC DMS is based on use of RC rescue medications (loratadine, olopatadine, mometasone), with different rescue medications being assigned different scores/dose unit (score range: 0-20). Lower DMS indicates less RC medication use. Summed RC DSS+DMS could range from 0 to 38; a lower score indicates less RC symptoms and medication use. Components that contribute to DSS and DMS endpoints are collected in an electronic diary (e-diary) completed by the participant/parent/guardian. Evaluation is based on average TCS during peak RS.
Time Frame: The 15-day period during the ragweed season with the highest moving pollen average
Population: The analysis population includes all treated participants w/ ≥1 e-diary entry for the specified measurement and timeframe.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Short Ragweed Pollen Allergen Extract | Placebo
Number analyzed (Participants) | 460 | 487
Score on a scale | 4.39 (3.85) [3.85 to 4.94] | 7.12 (6.57) [6.57 to 7.67]
Statistical Analysis 1: Comparison: Short Ragweed Pollen Allergen Extract vs Placebo; Test type: Superiority; p < 0.001, ANOVA; Model included fixed effects of treatment, baseline asthma status, age group, pollen season, and pollen region nested within pollen season; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-3.45 to -2.00]

2. Secondary Outcome: Average TCS During the Entire RS
Description: TCS is DSS plus DMS, assessed here during the entire RS. This starts from the first day of 3 consecutive days with ragweed pollen counts ≥10 grains/m^3 through the last day of the last occurrence of 3 consecutive days with ragweed pollen counts ≥10 grains/m^3. The duration of the entire RS is up to 13 weeks; this duration varies by site/region. The RC DSS assesses 6 allergy symptoms measured on a scale of 0 to 3 (score range: 0-18). A lower DSS indicates less RC symptoms. The RC DMS is based on use of RC rescue medications (loratadine, olopatadine, mometasone) with different scores/dose unit (score range: 0-20). A lower DMS indicates less RC medication use. The sum of RC DSS+DMS ranges from 0 to 38, with a lower score indicating less RC symptoms and medication use. Components contributing to the TCS for the entire RS are collected in an e-diary completed by the participant/parent/guardian.
Time Frame: Up to 13 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Short Ragweed Pollen Allergen Extract | Placebo
Number analyzed (Participants) | 466 | 491
Score on a scale | 3.88 (3.44) [3.44 to 4.33] | 5.75 (5.30) [5.30 to 6.20]
Statistical Analysis 1: Comparison: Short Ragweed Pollen Allergen Extract vs Placebo; Test type: Superiority; p < 0.001, ANOVA; [statistical method as in outcome 1, analysis 1]; Difference in LS Mean = -1.86, 95% CI 2-sided [-2.46 to -1.27]

3. Secondary Outcome: Average Rhinoconjunctivitis (RC) DSS During the Peak RS
Description: The DSS consists of a total of 6 rhinoconjunctivitis symptoms: 4 rhinitis symptoms (runny nose, stuffy nose, sneezing, itchy nose) and 2 conjunctivitis symptoms (itchy eyes, watery eyes). The components that contribute to the DSS endpoint are collected in an e-diary completed by the participant/parent/guardian. The RC DSS is measured on a 4-point scale from 0 to 3 as follows: 0 (no sign/symptom evident) to 3 (sign/symptom that is hard to tolerate; may cause interference with activities of daily living and/or sleeping). The maximum DSS is 18 points if a participant experiences all 6 symptoms with an intensity of 3 for each symptom. The minimum DSS is 0 points if a participant experiences no symptoms. A lower DSS means symptoms are less severe. The evaluation is based on the average DSS during the peak RS.
Time Frame: The 15-day period during the ragweed season with the highest moving pollen average
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Short Ragweed Pollen Allergen Extract | Placebo
Number analyzed (Participants) | 468 | 494
Score on a scale | 2.55 (2.24) [2.24 to 2.86] | 3.95 (3.63) [3.63 to 4.26]
Statistical Analysis 1: Comparison: Short Ragweed Pollen Allergen Extract vs Placebo; Test type: Superiority; p < 0.001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.40, 95% CI 2-sided [-1.81 to -0.99]

4. Secondary Outcome: Average Rhinoconjunctivitis (RC) DMS During the Peak RS
Description: This DMS endpoint consists of a total of scores for use of RC medications: loratadine syrup or tablets (6 points), olopatadine (6 points), and mometasone (8 points). The score range of the RC DMS is 0-20 points, and a lower DMS means that less medication is used. The method used for analysis of the RC DMS is a zero-inflated log-normal model, which takes the average RC DMS during the peak RS as the response and adjusts for the same terms as in the ANOVA model. The components that contribute to the DMS endpoint are collected in an e-diary completed by the participant/parent/guardian.
Time Frame: The 15-day period during the ragweed season with the highest moving pollen average
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Short Ragweed Pollen Allergen Extract | Placebo
Number analyzed (Participants) | 460 | 487
Score on a scale | 2.01 (1.57) [1.57 to 2.46] | 3.85 (3.14) [3.14 to 4.57]
Statistical Analysis 1: Comparison: Short Ragweed Pollen Allergen Extract vs Placebo; Test type: Superiority; p < 0.001, Zero-Inflated Log-Normal Model; Model included fixed effects of treatment, baseline asthma, age group, pollen season, and pollen region nested within pollen season; Mean Difference (Final Values) = -1.84, 95% CI 2-sided [-2.60 to -1.08]

5. Secondary Outcome: Percentage of Participants Reporting Pre-specified Local Application Site Reactions
Description: Pre-specified local application site reactions, irrespective of causality, included AEs related to lip swelling/edema, mouth swelling/edema, palatal swelling/edema, swollen tongue/edema, oropharyngeal swelling/edema, pharyngeal edema/throat tightness, oral pruritus, throat irritation, tongue pruritus, and ear pruritus.
Time Frame: Up to 35 weeks
Population: The safety population was all participants as treated. One participant was randomized to placebo but received short ragweed pollen allergen extract for one day and is included in the short ragweed pollen allergen extract arm.
Measure: Number; unit: Percentage of Participants
Groups:
- Short Ragween Pollen Allergen Extract: Participants received one short ragweed pollen allergen extract sublingual tablet containing 12 units of Amb a 1-U, QD for up to 35 weeks.
Arm/Group | Short Ragween Pollen Allergen Extract | Placebo
Number analyzed (Participants) | 513 | 509
Percentage of Participants | 64.52 | 26.92
Statistical Analysis 1: Comparison: Short Ragween Pollen Allergen Extract vs Placebo; Test type: Other; p < 0.001, Miettinen & Nurminen; Difference in % estimates = 37.61, 95% CI 2-sided [31.82 to 43.12]

6. Secondary Outcome: Percentage of Participants Reporting Anaphylaxis and/or Systemic Allergic Reactions
Description: For the purposes of this study, systemic allergic reactions are allergic reactions that occur away from the site of study drug application (allergic reactions other than local application site reactions). Anaphylaxis is a severe allergic reaction that typically involves more than one body system.
Time Frame: Up to 35 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Short Ragweed Pollen Allergen Extract | Placebo
Number analyzed (Participants) | 513 | 509
Percentage of Participants | 0.58 | 0.20
Statistical Analysis 1: Comparison: Short Ragweed Pollen Allergen Extract vs Placebo; Test type: Other; p = 0.320, Miettinen & Nurminen; Difference in % estimates = 0.39, 95% CI 2-sided [-0.57 to 1.53]

7. Secondary Outcome: Percentage of Participants Treated With Epinephrine
Description: Self-injectable epinephrine was provided to each participant/parent/guardian at randomization in countries where it is a regulatory requirement, and was to be available around the time treatment is administered at home. Self-injectable epinephrine was intended for immediate self-administration for an anaphylactic reaction, including symptoms/signs of upper airway obstruction. Instances of treatment with forms of epinephrine other than systemic epinephrine (e.g., inhaled racepinephrine) were counted as use of epinephrine.
Time Frame: Up to 35 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Short Ragween Pollen Allergen Extract | Placebo
Number analyzed (Participants) | 513 | 509
Percentage of Participants | 0.19 | 0.20
Statistical Analysis 1: Comparison: Short Ragween Pollen Allergen Extract vs Placebo; Test type: Other; p = 0.996, Miettinen & Nurminen; Difference in % estimates = 0.00, 95% CI 2-sided [-0.92 to 0.92]

ADVERSE EVENTS:
Time Frame: Up to 35 weeks
Description: An AE is any physical or clinical change or disease experienced by the participant at any time during the course of the study, whether or not considered related to the use of the study drug. The safety population was all participants as treated. One participant was randomized to placebo but received short ragweed pollen allergen extract for one day and is included in the short ragweed pollen allergen extract arm.
Arm/Group | Short Ragweed Pollen Allergen Extract | Placebo
All-Cause Mortality (participants affected / at risk) | 0/513 | 0/509
Serious Adverse Events (participants affected / at risk) | 7/513 | 9/509
Other Adverse Events (participants affected / at risk) | 370/513 | 233/509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Ragweed Pollen Allergen Extract (N=513) | Placebo (N=509)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Conduct disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal viral inection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Ragweed Pollen Allergen Extract (N=513) | Placebo (N=509)
Ear pruritus (Ear and labyrinth disorders) | 177 (750) | 35 (65)
Abdominal pain upper (Gastrointestinal disorders) | 54 (119) | 30 (53)
Diarrhoea (Gastrointestinal disorders) | 26 (55) | 21 (29)
Enlarged uvula (Gastrointestinal disorders) | 33 (65) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 64 (171) | 13 (29)
Lip swelling (Gastrointestinal disorders) | 66 (165) | 7 (14)
Nausea (Gastrointestinal disorders) | 70 (167) | 43 (69)
Oral pain (Gastrointestinal disorders) | 64 (151) | 16 (29)
Oral pruritus (Gastrointestinal disorders) | 247 (1115) | 62 (131)
Stomatitis (Gastrointestinal disorders) | 34 (89) | 6 (13)
Swollen tongue (Gastrointestinal disorders) | 56 (132) | 4 (5)
Pyrexia (General disorders) | 29 (33) | 20 (23)
Nasopharyngitis (Infections and infestations) | 38 (50) | 36 (50)
Headache (Nervous system disorders) | 45 (100) | 49 (67)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (39) | 30 (53)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 (56) | 29 (44)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 58 (138) | 8 (14)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 254 (1048) | 98 (223)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (2):
  • Study Protocol (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT02478398/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT02478398/SAP_001.pdf